CLINICAL TRIAL: NCT02170181
Title: UTSW SBRT Prospective Clinical Registry for Oligometastic Disease, Consolidation Therapy, Debulking Prior to Chemotherapy, or Re-Irradiation
Brief Title: Clinical Registry for Oligometastic Disease, Consolidation Therapy, Debulking Prior to Chemotherapy, or Re-Irradiation
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Asal Rahimi, Associate Professor of Medicine, University of Texas Southwestern Medical Center
Other Study IDs: STU 012014-039
Record Dates: First submitted 2014-06-13; First posted 2014-06-23 (Estimated); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Cancer Patients Receiving Stereotactic Body RTX
Keywords: SBRT; prostate cancer; lung cancer; bladder cancer; kidney cancer; oligometastatic disease
MeSH Terms: conditions — Prostatic Neoplasms; Lung Neoplasms; Urinary Bladder Neoplasms; Kidney Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Tissue Procurement
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- OLIGOMETASTATIC ARM: SBRT to Oligometastases
  Interventions: Radiation: SBRT
- CONSOLIDATION ARM: SBRT as Consolidation to Residual Disease
  Interventions: Radiation: SBRT
- NORTON-SIMON ARM: SBRT to Debulk Gross Disease
  Interventions: Radiation: SBRT
- RE-IRRADIATION ARM
  Interventions: Radiation: SBRT

INTERVENTIONS:
Radiation: SBRT — SBRT to Oligometastases
  Other Names: Stereotactic body radiation therapy

SUMMARY:
This prospective protocol will enroll patients with pathologically confirmed solid malignancies who receive stereotactic body radiation therapy (SBRT) for oligometastases, for consolidation after systemic therapy, prior to systemic therapy for the purposes of debulking, or in the re-irradiation setting. Increasing use of SBRT off of clinical trials in patients with malignancies of all histologies is being utilized in these settings. However, individualized outcomes and characteristics of treatments are not prospectively followed and not well documented. By instituting a registry of patients receiving SBRT in these settings it will be possible to determine trends in patterns of care and outcomes for refinement and justification of this treatment.

DETAILED DESCRIPTION:
Patients will be grouped into one of four treatment arms. Treatment intent must be specified at the time of registration.

OLIGOMETASTATIC ARM- The first treatment arm will be for patients with oligometastatic disease, which will be defined as a treatment with curative intent to less than or equal to six sites of disease on initial presentation of metastatic disease or within the context of the initial combined modality treatment regimen (e.g., after a chemotherapy or surgical phase of therapy). Patients in this treatment arm will receive a definitive, ablative dose of radiation intended to eradicate all residual gross tumor of "all" sites of disease. A variety of acceptable ablative fractionation schemes with variable ability to prevent normal tissue toxicity will be allowed. Further planned systemic therapy or surgery does not eliminate stratification into this group so long as the overall intent is curative.

CONSOLIDATION ARM- The second treatment arm will be for consolidation following systemic therapy. This approach is akin to the experience with consolidation with radiation with conventional radiation after systemic therapy for tumors like bulky lymphomas, etc. In this context, treatment will be directed towards PET-avid residual disease assuming them to harbor residual active disease or disease more resistant to systemic therapy. The treatment doses will be sub-ablative yet will still maintain radiobiologic potency for local control with the option in the future for further systemic therapy.

NORTON-SIMON ARM- The third treatment arm will enroll patients prior to receiving systemic therapy who require initial debulking of gross disease to enhance chemotherapy efficacy per the Norton-Simon hypothesis. (Patients who initially receive systemic therapy, with gross residual disease in less than or equal to 6 sites of disease, who then receive SBRT with planned further systemic therapy (targeted or cytotoxic) immediately following SBRT will be enrolled onto this arm)

RE-IRRADIATION ARM- The fourth treatment arm will enroll patients if they have had prior irradiation and suffered disease recurrence or failure within a previously irradiated volume. Prior irradiation can consist of external beam irradiation- conventional treatment, hypofractionated treatment, stereotactic radiation, or even brachytherapy

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed solid tumor malignancies which are locally advanced or metastatic.
2. Able to safely receive intended protocol defined SBRT dose.
3. For oligometastatic category, patients can have up to 6 sites of active extracranial disease amenable to SBRT with a maximum of 7 cm diameter
4. Must have a CT C/A/P, or PET/CT scan within 12 weeks of enrollment.
5. Age ≥ 18 years.
6. Karnofsky performance status of 70 or higher, or ECOG < 2
7. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

   7.1 a female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:
   * Has not undergone a hysterectomy or bilateral oophorectomy; or
   * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
8. Negative urine or serum pregnancy test for women of child-bearing potential
9. Agreeable and willing to participate in expected protocol defined follow-up.
10. Ability to understand and the willingness to sign a written informed consent.
11. Registry participation does not exclude participation in clinical trials.

Exclusion Criteria:

1 Because the tolerance dose of SBRT to the gastrointestinal tract is not established, patients with metastatic disease invading the esophagus, stomach, intestines, or mesenteric lymph nodes will not be eligible.

2. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

3 Subjects must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients receive SBRT
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2014-05-28 (Actual); Primary Completion 2025-08 (Actual); Study Completion 2025-08 (Actual)

PRIMARY OUTCOMES:
patterns of care | 5 years
  Prospectively enroll patients to one of four treatment categories who are to receive SBRT onto a registry to define patterns of care:
  Group 1: Oligometastatic disease- all radiologic suspicious areas for viable disease to be treated
  Group 2: Consolidation Therapy - only PET avid or progressive disease
  Group 3: Norton-Simon Arm - SBRT prior to initial of planned further systemic therapy
  Group 4: Re-Irradiation Arm-recurrence or failure within a previously irradiated volume.

SECONDARY OUTCOMES:
Loco-regional control | 5 years
  Loco-regional control in sites treated via SBRT in the four treatment categories.
overall survival | 5 years
  To evaluate overall survival among patients in the four treatment categories.
Number of patients with toxicities | 5 years
  To evaluate the safety of SBRT in the four treatment categories: toxicities review

CONTACTS AND LOCATIONS:
Overall Officials: Asal Rahimi, MD, Principal Investigator — UTSW
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States